CLINICAL TRIAL: NCT02559895
Title: A Parallel Group, Double-Blind, Randomized, Placebo Controlled, Trial to Evaluate the Efficacy and Safety of ALD403 Administered Intravenously in Patients With Frequent Episodic Migraines
Brief Title: A Multicenter Assessment of ALD403 in Frequent Episodic Migraine
Acronym: PROMISE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alder Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ALD403-CLIN-006
Record Dates: First submitted 2015-09-22; First posted 2015-09-25 (Estimated); Results first posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — eptinezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ALD403 Dose Level 1 (Experimental): ALD403 Dose Level 1 (IV)
  Interventions: Drug: ALD403
- ALD403 Dose Level 2 (Experimental): ALD403 Dose Level 2 (IV)
  Interventions: Drug: ALD403
- ALD403 Dose Level 3 (Experimental): ALD403 Dose Level 3 (IV)
  Interventions: Drug: ALD403
- Placebo (Placebo Comparator): Placebo (IV)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALD403
  Other Names: Eptinezumab-jjmr; Vyepti
  Arms: ALD403 Dose Level 1; ALD403 Dose Level 2; ALD403 Dose Level 3
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess ALD403 in the prevention of migraine headache in frequent episodic migraineurs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine at ≤ 50 years of age (ICHD-II, 2004 Section 1)
* History of migraine ≥ 12 months with

  * ≤ 14 headache days of which at least 4 have to be migraine days (migraine days count as headache days) in each 28 day period in the 3 months prior to screening
  * During the 28 days following the screening visit, the subject experiences ≤ 14 headache days of which at least 4 have to be migraine days (migraine days count as headache days) as recorded in the eDiary
* No use of any botulinum toxin for migraine or for any other medical/cosmetic reasons requiring injections in the head, face, or neck 4 months prior to screening and during the 28 day period prior to randomization
* Headache eDiary was completed on at least 25 of the 28 days prior to randomization

Exclusion Criteria:

* Confounding pain syndromes, e.g. fibromyalgia, complex regional pain syndrome or any pain syndrome that requires regular analgesia
* Psychiatric conditions that are uncontrolled and untreated, including conditions that are not controlled for a minimum of 6 months prior to screening
* History or diagnosis of complicated migraine (ICHD- II, 2004 Section 1), chronic tension-type headache, hypnic headache, cluster headache, hemicrania continua, new daily persistent headache, migraine with brainstem aura, sporadic and familial hemiplegic migraine
* Unable to differentiate migraine from other headaches
* Have any clinically significant concurrent medical condition
* Receipt of any monoclonal antibody treatment within 6 months of screening (within or outside a clinical trial)
* Previously dosed with ALD403 or any monoclonal antibody targeting the CGRP pathway

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 898 (Actual)
Dates: Start 2015-09; Primary Completion 2017-02 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Whitaker, MD, Study Director — Alder Biopharmaceuticals, Inc.
Locations (77):
- United States (76):
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Fresno, California
  - Research Site, Fullerton, California
  - Research Site, Long Beach, California
  - Research Site, Montclair, California
  - Research Site, Oceanside, California
  - Research Site, Redlands, California
  - Research Site, San Diego, California
  - Research Site, Santa Monica, California
  - Research Site, Sherman Oaks, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Fort Collins, Colorado
  - Research Site, Stamford, Connecticut
  - Research Site, Waterbury, Connecticut
  - Research Site, Bradenton, Florida
  - Research Site, DeLand, Florida
  - Research site, Fort Myers, Florida
  - Research Site, Hallandale, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Maitland, Florida
  - Research Site, Miami, Florida
  - Research Site, Naples, Florida
  - Research Site, Orlando, Florida
  - Research Site, Sunrise, Florida
  - Research Site, Winter Haven, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Stockbridge, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Lisle, Illinois
  - Research Site, Prairie Village, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Owensboro, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Boston, Massachusetts
  - Research Site, North Attleboro, Massachusetts
  - Research Site, Springfield, Massachusetts
  - Research Site, Watertown, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Farmington Hills, Michigan
  - Research Site, Jackson, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Flowood, Mississippi
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Albuquerque, New Mexico
  - Research Site, Brooklyn, New York
  - Research Site, Hartsdale, New York
  - Research Site, Rochester, New York
  - Research Site, Staten Island, New York
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Dayton, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Norman, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Allentown, Pennsylvania
  - Research Site, Smithfield, Pennsylvania
  - Research Site, Anderson, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Kingsport, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Bellevue, Washington
- Research Site, Tbilisi, Georgia

REFERENCES:
- [Derived] Pozo-Rosich P, Dodick DW, Ettrup A, Hirman J, Cady R. Shift in diagnostic classification of migraine after initiation of preventive treatment with eptinezumab: post hoc analysis of the PROMISE studies. BMC Neurol. 2022 Oct 25;22(1):394. doi: 10.1186/s12883-022-02914-9. PMID 36284281
- [Derived] Apelian R, Boyle L, Hirman J, Asher D. Measuring dose-related efficacy of eptinezumab for migraine prevention: post hoc analysis of PROMISE-1 and PROMISE-2. J Headache Pain. 2022 Apr 18;23(1):48. doi: 10.1186/s10194-022-01418-8. PMID 35436857
- [Derived] Ashina M, McAllister P, Cady R, Hirman J, Ettrup A. Efficacy and safety of eptinezumab in patients with migraine and self-reported aura: Post hoc analysis of PROMISE-1 and PROMISE-2. Cephalalgia. 2022 Jul;42(8):696-704. doi: 10.1177/03331024221077646. Epub 2022 Mar 18. PMID 35302389
- [Derived] Martin V, Nagy AJ, Janelidze M, Giorgadze G, Hirman J, Cady R, Mehta L, Buse DC. Impact of Baseline Characteristics on the Efficacy and Safety of Eptinezumab in Patients With Migraine: Subgroup Analyses of PROMISE-1 and PROMISE-2. Clin Ther. 2022 Mar;44(3):389-402. doi: 10.1016/j.clinthera.2022.01.006. Epub 2022 Feb 5. PMID 35131090
- [Derived] Lipton RB, Charleston L 4th, Tassorelli C, Brevig T, Hirman J, Cady R. Patient-reported outcomes, health-related quality of life, and acute medication use in patients with a >/= 75% response to eptinezumab: subgroup pooled analysis of the PROMISE trials. J Headache Pain. 2022 Feb 7;23(1):23. doi: 10.1186/s10194-022-01386-z. PMID 35130836
- [Derived] Smith TR, Spierings ELH, Cady R, Hirman J, Ettrup A, Shen V. Cardiovascular outcomes in adults with migraine treated with eptinezumab for migraine prevention: pooled data from four randomized, double-blind, placebo-controlled studies. J Headache Pain. 2021 Nov 25;22(1):143. doi: 10.1186/s10194-021-01360-1. PMID 34823467
- [Derived] Smith TR, Spierings ELH, Cady R, Hirman J, Schaeffler B, Shen V, Sperling B, Brevig T, Josiassen MK, Brunner E, Honeywell L, Mehta L. Safety and tolerability of eptinezumab in patients with migraine: a pooled analysis of 5 clinical trials. J Headache Pain. 2021 Mar 30;22(1):16. doi: 10.1186/s10194-021-01227-5. PMID 33781209
- [Derived] Smith TR, Janelidze M, Chakhava G, Cady R, Hirman J, Allan B, Pederson S, Smith J, Schaeffler B. Eptinezumab for the Prevention of Episodic Migraine: Sustained Effect Through 1 Year of Treatment in the PROMISE-1 Study. Clin Ther. 2020 Dec;42(12):2254-2265.e3. doi: 10.1016/j.clinthera.2020.11.007. Epub 2020 Nov 27. PMID 33250209
- [Derived] Ashina M, Saper J, Cady R, Schaeffler BA, Biondi DM, Hirman J, Pederson S, Allan B, Smith J. Eptinezumab in episodic migraine: A randomized, double-blind, placebo-controlled study (PROMISE-1). Cephalalgia. 2020 Mar;40(3):241-254. doi: 10.1177/0333102420905132. Epub 2020 Feb 19. PMID 32075406

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 2413 participants signed the ICF, of which 898 participants met the entry criteria and were randomized into the trial.
Groups:
- 300 mg ALD403: Participants were randomized to receive a single 300 mg IV infusion of ALD403 on Days 0, 84 (Week 12), 168 (Week 24) and 252 (Week 36).
- 100 mg ALD403: Participants were randomized to receive a single 100 mg IV infusion of ALD403 on Days 0, 84 (Week 12), 168 (Week 24) and 252 (Week 36).
- 30 mg ALD403: Participants were randomized to receive a single 30 mg IV infusion of ALD403 on Days 0, 84 (Week 12), 168 (Week 24) and 252 (Week 36).
- Placebo: Participants were randomized to receive a single placebo IV infusion on Days 0, 84 (Week 12), 168 (Week 24) and 252 (Week 36).
Period: Overall Study
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo
Started | 224 | 225 | 224 | 225
Participants Treated (2 participants received duplicate randomization, participants are summarized in first group assigned) | 222 | 221 | 223 | 222
Completed | 169 | 172 | 170 | 165
Not Completed | 55 | 53 | 54 | 60
Not completed — Adverse Event | 3 | 3 | 2 | 1
Not completed — Lack of Efficacy | 2 | 3 | 2 | 8
Not completed — Lost to Follow-up | 22 | 16 | 12 | 17
Not completed — Physician Decision | 1 | 1 | 3 | 0
Not completed — Withdrawal by Subject | 16 | 9 | 20 | 9
Not completed — Study Burden | 10 | 16 | 12 | 22
Not completed — Other | 1 | 5 | 3 | 3

BASELINE CHARACTERISTICS:
Population: Safety population includes all participants who received study drug or placebo. 2 participants received duplicate randomization, participants are summarized within treatment group for which they actually received treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo | Total
Number analyzed (Participants) | 224 | 223 | 219 | 222 | 888
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (11.72) | 40.0 (10.66) | 39.1 (11.54) | 39.9 (11.67) | 39.8 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199 | 179 | 185 | 186 | 749
  Male | 25 | 44 | 34 | 36 | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 42 | 45 | 34 | 161
  Not Hispanic or Latino | 184 | 181 | 174 | 188 | 727
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 1 | 3
  Asian | 1 | 1 | 1 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 1 | 3
  Black or African American | 27 | 17 | 31 | 30 | 105
  White | 187 | 196 | 180 | 181 | 744
  More than one race | 5 | 7 | 5 | 5 | 22
  Unknown or Not Reported | 1 | 1 | 2 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 185 | 184 | 194 | 185 | 748
  Georgia | 39 | 39 | 25 | 37 | 140
Number of migraine days [Mean (Standard Deviation); unit: Days] — Self reported average number of migraine days per 28-day period in the 3 months prior to screening.
  Days | 7.8 (2.59) | 7.5 (2.60) | 7.9 (2.70) | 7.5 (2.42) | 7.7 (2.58)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Monthly Migraine Days (Weeks 1-12)
Description: Monthly migraine days are summarized in 28-day intervals, and averaged across Weeks 1-12
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Mean (Standard Deviation); unit: Migraine Days
Groups:
- 300 mg ALD403: Participants received a single 300 mg IV infusion of ALD403 on Days 0, 84 (Week 12), 168 (Week 24) and 252 (Week 36).
- 100 mg ALD403: Participants received a single 100 mg IV infusion of ALD403 on Days 0, 84 (Week 12), 168 (Week 24) and 252 (Week 36).
- 30 mg ALD403: Participants received a single 30 mg IV infusion of ALD403 on Days 0, 84 (Week 12), 168 (Week 24) and 252 (Week 36).
- Placebo: Participants received a single placebo IV infusion on Days 0, 84 (Week 12), 168 (Week 24) and 252 (Week 36).
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo
Number analyzed (Participants) | 222 | 221 | 223 | 222
Migraine Days | -4.3 (3.42) | -3.9 (3.23) | -4.1 (3.22) | -3.1 (3.70)
Statistical Analysis 1: Comparison: 300 mg ALD403 vs Placebo; Test type: Superiority; p = 0.0001, ANCOVA; Mean Difference (Final Values) = -1.11, 95% CI 2-sided [-1.68 to -0.54], Standard Deviation 3.40
Statistical Analysis 2: Comparison: 100 mg ALD403 vs Placebo; Test type: Superiority; p = 0.0182, ANCOVA; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-1.25 to -0.12], Standard Deviation 3.40
Statistical Analysis 3: Comparison: 30 mg ALD403 vs Placebo; Test type: Superiority; p = 0.0046, ANCOVA; Mean Difference (Final Values) = -0.82, 95% CI 2-sided [-1.39 to -0.25], Standard Deviation 3.40

2. Secondary Outcome: 75% Migraine Responder Rate
Description: Participants with an average reduction in migraine days of at least 75% over Weeks 1 to 12, as compared with baseline.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo
Number analyzed (Participants) | 222 | 221 | 223 | 222
Participants | 66 | 49 | 55 | 36
Statistical Analysis 1: Comparison: 300 mg ALD403 vs Placebo; Test type: Superiority; p = 0.0007, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 13.5, 95% CI 2-sided [5.8 to 21.2]
Statistical Analysis 2: Comparison: 100 mg ALD403 vs Placebo; Test type: Superiority; p = 0.1126, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 6.0, 95% CI 2-sided [-1.4 to 13.3]
Statistical Analysis 3: Comparison: 30 mg ALD403 vs Placebo; Test type: Superiority; p = 0.0272, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 8.4, 95% CI 2-sided [1.0 to 15.9]

3. Secondary Outcome: 75% Migraine Responder Rate
Description: Participants with an average reduction in migraine days of at least 75% over Weeks 1 to 4, as compared with baseline.
Time Frame: Week 1-4
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo
Number analyzed (Participants) | 222 | 221 | 223 | 222
Participants | 70 | 68 | 67 | 45
Statistical Analysis 1: Comparison: 300 mg ALD403 vs Placebo; Test type: Superiority; p = 0.0066, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 11.3, 95% CI 2-sided [3.2 to 19.3]
Statistical Analysis 2: Comparison: 100 mg ALD403 vs Placebo; Test type: Superiority; p = 0.0112, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 10.5, 95% CI 2-sided [2.4 to 18.6]
Statistical Analysis 3: Comparison: 30 mg ALD403 vs Placebo; Test type: Superiority; p = 0.0170, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 9.8, 95% CI 2-sided [1.8 to 17.8]

4. Secondary Outcome: 50% Migraine Responder Rate
Description: Participants with an average reduction in migraine days of at least 50% over Weeks 1 to 12, as compared with baseline
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo
Number analyzed (Participants) | 222 | 221 | 223 | 222
Participants | 125 | 110 | 112 | 83
Statistical Analysis 1: Comparison: 300 mg ALD403 vs Placebo; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 18.9, 95% CI 2-sided [9.8 to 28.0]
Statistical Analysis 2: Comparison: 100 mg ALD403 vs Placebo; Test type: Superiority; p = 0.0085, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 12.4, 95% CI 2-sided [3.2 to 21.5]
Statistical Analysis 3: Comparison: 30 mg ALD403 vs Placebo; Test type: Superiority; p = 0.0064, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 12.8, 95% CI 2-sided [3.7 to 22.0]

5. Secondary Outcome: Percentage of Participants With a Migraine on the Day After Dosing
Description: The percentage of participants with a migraine on the day after dosing, where Day 0 is treatment day and Day 1 is the day after dosing
Time Frame: 1 day
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Number; unit: Percentage of participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo
Number analyzed (Participants) | 222 | 221 | 223 | 222
Percentage of participants | 13.9 | 14.8 | 17.3 | 22.5
Statistical Analysis 1: Comparison: 300 mg ALD403 vs Placebo; Test type: Superiority; p = 0.0159, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: 100 mg ALD403 vs Placebo; Test type: Superiority; p = 0.0312, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: 30 mg ALD403 vs Placebo; Test type: Superiority; p = 0.1539, Cochran-Mantel-Haenszel

6. Secondary Outcome: 75% Headache Responder Rate
Description: Participants with an average reduction in headache days of at least 75% over Weeks 1 to 12, as compared with baseline.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo
Number analyzed (Participants) | 222 | 221 | 223 | 222
Participants | 42 | 28 | 34 | 23

7. Secondary Outcome: 50% Headache Responder Rate
Description: Participants with an average reduction in headache days of at least 50% over Weeks 1 to 12, as compared with baseline.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo
Number analyzed (Participants) | 222 | 221 | 223 | 222
Participants | 113 | 98 | 98 | 74

8. Secondary Outcome: 100% Migraine Responder Rate
Description: Participants with a reduction in migraine days of 100% over Weeks 1 to 12, as compared with baseline
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo
Number analyzed (Participants) | 222 | 221 | 223 | 222
Participants | 9 | 1 | 4 | 4

9. Secondary Outcome: 100% Headache Responder Rate
Description: Participants with a reduction in headache days of 100% over Weeks 1 to 12, as compared with baseline.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo
Number analyzed (Participants) | 222 | 221 | 223 | 222
Participants | 6 | 0 | 4 | 2

10. Secondary Outcome: Change From Baseline in Acute Migraine Medication Days (Weeks 1-12)
Description: The change in number of days with any triptan or ergotamine use as recorded in the eDiary.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo
Number analyzed (Participants) | 222 | 221 | 223 | 222
days | -0.8 (1.77) | -0.9 (2.00) | -0.6 (1.62) | -0.4 (1.27)

11. Secondary Outcome: Change From Baseline in Average Daily Migraine Prevalence to Week 4
Description: The change in the percentage of days where a participant has a migraine from baseline to Week 4.
Time Frame: Baseline to Week 4
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Mean (Standard Deviation); unit: percentage of days with migraine
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo
Number analyzed (Participants) | 222 | 221 | 223 | 222
percentage of days with migraine | -14.9 (19.78) | -13.8 (19.27) | -15.1 (17.83) | -9.7 (19.33)

12. Secondary Outcome: Change From Baseline to Week 12 in Percentage of Migraines With Use of Acute Medication
Description: The percentage of migraines with acute medication usage. Participants with no migraines will be included with a rate of zero.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Mean (Standard Deviation); unit: percentage of acute medication migraines
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo
Number analyzed (Participants) | 222 | 221 | 223 | 222
percentage of acute medication migraines | 62.08 (38.46) | 66.58 (34.13) | 69.11 (33.72) | 71.44 (34.59)

13. Secondary Outcome: Change From Baseline to Week 12 in Percentage of Headaches With Use of Acute Medication
Description: The percentage of headaches with acute medication usage. Participants with no headaches will be included with a rate of zero.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Mean (Standard Deviation); unit: percentage of acute medication headaches
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo
Number analyzed (Participants) | 222 | 221 | 223 | 222
percentage of acute medication headaches | 63.09 (36.87) | 66.85 (33.65) | 67.84 (33.59) | 70.95 (33.43)

14. Secondary Outcome: Change From Baseline in Monthly Headache Days (Weeks 1-12)
Description: Monthly headache days are summarized in 28-day intervals, and averaged across Weeks 1-12.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Mean (Standard Deviation); unit: headache days
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo
Number analyzed (Participants) | 222 | 221 | 223 | 222
headache days | -4.5 (3.96) | -4.0 (3.30) | -4.4 (3.24) | -3.3 (3.51)

15. Secondary Outcome: Percent of Headaches With Severe Intensity
Description: Summary of percent of headaches with severe intensity over Weeks 1-12.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Mean (Standard Deviation); unit: percentage of severe intensity headaches
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo
Number analyzed (Participants) | 222 | 221 | 223 | 222
percentage of severe intensity headaches | 17.06 (22.03) | 19.84 (24.83) | 21.20 (26.60) | 21.68 (22.67)

16. Secondary Outcome: Percent of Migraines With Severe Intensity
Description: Summary of percent of migraines with severe intensity over Week 1-12.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Mean (Standard Deviation); unit: percentage of severe intensity migraines
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo
Number analyzed (Participants) | 222 | 221 | 223 | 222
percentage of severe intensity migraines | 19.07 (23.46) | 22.23 (26.30) | 24.43 (28.15) | 26.01 (24.99)

17. Secondary Outcome: Change From Baseline in Monthly Migraine Hours (Weeks 1-12)
Description: Migraine hours are the sum of the duration of migraines within 4 week intervals, and the average 4 week duration within 12 week intervals.
Time Frame: Week 1-12
Measure: Mean (Standard Deviation); unit: migraine hours
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo
Number analyzed (Participants) | 222 | 221 | 223 | 222
migraine hours | -42.9 (49.91) | -35.3 (47.85) | -37.8 (50.17) | -23.8 (50.91)

18. Secondary Outcome: Change From Baseline in Monthly Headache Hours, Weeks 1-12
Description: Headache hours are the sum of the duration of headaches within 4 week intervals, and the average 4 week duration within 12 week intervals.
Time Frame: Week 1-12
Measure: Mean (Standard Deviation); unit: headache hours
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo
Number analyzed (Participants) | 222 | 221 | 223 | 222
headache hours | -42.0 (56.67) | -34.2 (49.19) | -38.8 (50.45) | -24.5 (48.15)

19. Secondary Outcome: Change From Baseline of Short Form Health Survey (SF-36 v 2.0) Scale Scores
Description: The SF-36 is a health survey containing 36 questions consisting of eight scaled scores to measure quality of life over the past 4 weeks. All scales are on a range of 0 to 100, with 0 being the worst and 100 being the best. Scales are reported separately. Increases from baseline indicate improvement.
Time Frame: Baseline to Week 12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo. The Week 12 scores only include participants who completed the Week 12 visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo
Number analyzed (Participants) | 211 | 208 | 205 | 201
score on a scale
  Physical Functioning | 0.9 (5.78) | 1.2 (6.88) | 0.9 (6.74) | 0.3 (6.43)
  Role Physical | 3.0 (6.54) | 2.3 (7.65) | 2.4 (7.72) | 2.2 (6.78)
  Bodily Pain | 4.5 (8.27) | 4.3 (8.37) | 3.5 (9.12) | 2.3 (8.70)
  General Health | 1.2 (6.78) | 0.7 (7.22) | 0.6 (7.54) | 0.0 (6.52)
  Vitality | 2.3 (7.91) | 1.8 (8.36) | 0.2 (8.61) | 1.7 (7.43)

20. Secondary Outcome: Health Related Quality of Life (EQ-5D-5L) at Week 12
Description: The EQ-5D-5L is a descriptive system of health-related quality of life states consisting of 5 dimension/questions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of five responses. The responses record five levels of severity (no problems/slight problems/moderate problems/severe problems/extreme problems) within a particular EQ-5D dimension.
Time Frame: Week 12
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo
Number analyzed (Participants) | 208 | 206 | 201 | 198
Participants
  Mobility: No problems | 183 | 181 | 181 | 179
  Mobility: Slight problems | 21 | 18 | 16 | 15
  Mobility: Moderate problems | 4 | 6 | 3 | 4
  Mobility: Severe problems | 0 | 1 | 1 | 0
  Mobility: Extreme problems | 0 | 0 | 0 | 0
  Self-care: No problems | 206 | 201 | 198 | 195
  Self-care: Slight problems | 2 | 4 | 3 | 3
  Self-care: Moderate problems | 0 | 1 | 0 | 0
  Self-care: Severe problems | 0 | 0 | 0 | 0
  Self-care: Extreme problems | 0 | 0 | 0 | 0
  Usual Activities: No problems | 177 | 173 | 176 | 172
  Usual Activities: Slight problems | 29 | 22 | 21 | 19
  Usual Activities: Moderate problems | 2 | 10 | 3 | 7
  Usual Activities: Severe problems | 0 | 0 | 1 | 0
  Usual Activities: Extreme problems | 0 | 1 | 0 | 0
  Pain/Discomfort: No problems | 113 | 116 | 123 | 110
  Pain/Discomfort: Slight problems | 75 | 65 | 57 | 68
  Pain/Discomfort: Moderate problems | 19 | 24 | 18 | 18
  Pain/Discomfort: Severe problems | 1 | 1 | 3 | 2
  Pain/Discomfort: Extreme problems | 0 | 0 | 0 | 0
  Anxiety/Depression: No problems | 158 | 156 | 168 | 151
  Anxiety/Depression: Slight problems | 46 | 38 | 24 | 38
  Anxiety/Depression: Moderate problems | 3 | 9 | 8 | 8
  Anxiety/Depression: Severe problems | 1 | 2 | 0 | 0
  Anxiety/Depression: Extreme problems | 0 | 1 | 1 | 1

21. Secondary Outcome: Change in Baseline of Allodynia Symptom Checklist-12 (ASC-12) Total Score
Description: The ASC-12 includes 12 questions about the frequency of various allodynia symptoms in association with headache attacks. For individuals with more than one type of headache, questions are directed to the "most severe type of headache." Each item is measured in a Likert type scale option with response categories: "Does not apply to me", "never", "rarely", "less than half the time", and "half the time or more". ASC items were scored as 0 (i.e., never, rarely or does not apply to me), 1 (less than half the time), and 2 (half the time or more), yielding scores that ranged from 0 to 24. If a single item is missing, it is scored as a 0. If more than one item is missing the total score will be missing. The interpretation of the total score is, 0-2: none; 3-5: mild; 6-8: moderate; greater than or equal to 9: severe.
Time Frame: Baseline to Week 12
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo
Number analyzed (Participants) | 208 | 206 | 200 | 198
score on a scale | -1.6 (4.22) | -1.8 (3.90) | -1.6 (3.95) | -1.7 (4.33)

ADVERSE EVENTS:
Time Frame: Baseline to Week 56 (end of study)
Description: 2 participants received duplicate randomization, participants are summarized within treatment group for which they actually received treatment.
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/224 | 0/223 | 0/219 | 0/222
Serious Adverse Events (participants affected / at risk) | 3/224 | 4/223 | 4/219 | 6/222
Other Adverse Events (participants affected / at risk) | 44/224 | 44/223 | 44/219 | 41/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 300 mg ALD403 (N=224) | 100 mg ALD403 (N=223) | 30 mg ALD403 (N=219) | Placebo (N=222)
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic Cholestatic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Abdominal Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Postprocedural Complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Stomal Hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Benign Breast Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast Cancer Stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Panic Attack (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Uterine Prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Postprocedural Constipation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 300 mg ALD403 (N=224) | 100 mg ALD403 (N=223) | 30 mg ALD403 (N=219) | Placebo (N=222)
Nasopharyngitis (Infections and infestations) | 14 | 17 | 14 | 12
Sinusitis (Infections and infestations) | 11 | 6 | 7 | 14
Upper respiratory tract infection (Infections and infestations) | 23 | 22 | 25 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-04-24): https://cdn.clinicaltrials.gov/large-docs/95/NCT02559895/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/95/NCT02559895/SAP_001.pdf